CLINICAL TRIAL: NCT00652977
Title: Modified Ritgens Maneuver for Perineal Protection at Delivery
Brief Title: Ritgens Maneuver for the Prevention of Anal Sphincter Tears at Delivery: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Andreas Herbst, associate professor, Department of Obstetrics and Gynecology, Lund University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Lu1-99
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Last update posted 2008-04-07 (Estimated); Status verified 2008-04

CONDITIONS: Perineal Lacerations
Keywords: sphincter tears; Ritgen maneuver; perineal tears; prevention; delivery
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Active Comparator): The delivery of the fetal head should be managed by Ritgens maneuver, i.e. lifting the fetal chin anteriorly, using the fingers of one hand placed between the anus and the coccyx, and thereby extending the fetal neck, whereas the other hand should be placed on the fetal occiput to control the pace of the expulsion of the fetal head.
  Interventions: Procedure: Ritgens maneuver
- II (Other): Standard care at delivery: Manual support of the perineum
  Interventions: Procedure: Standard care (Manual support of the perineum)

INTERVENTIONS:
Procedure: Ritgens maneuver — Delivery of the fetal head should be managed by Ritgens maneuver, i.e. lifting the fetal chin anteriorly, using the fingers of one hand placed between the anus and the coccyx, and thereby extending the fetal neck, whereas the other hand should be placed on the fetal occiput to control the pace of the expulsion of the fetal head. The maneuver was used during a uterine contraction
  Arms: I
Procedure: Standard care (Manual support of the perineum) — The protocol entailed our standard care: using one hand to apply pressure against the perineum, and the other hand on the fetal occiput to control the expulsion of the fetal head, and only to use Ritgen´s maneuver in case of labor arrest or abnormal fetal heart rate pattern when the fetal head was at the pelvic floor.
  Arms: II

SUMMARY:
The aim of the investigation was to assess whether routine use of the modified Ritgen´s maneuver decreases the risk of anal sphincter injury at delivery, compared with simple manual protection of the perineum.Ritgen´s maneuver means that the fetal chin is reached for between the anus and the coccyx and pulled anteriorly, while using the fingers of the other hand on the fetal occiput to control speed of delivery and keep flexion of the fetal neck.

DETAILED DESCRIPTION:
This application is made retroactively - the study was performed during December 1st, 1999 to July 31st, 2001, at Lund University Hospital and Helsingborg Hospital. Primigravid women in the area were informed about the study at the maternity care centers, receiving written information in gestational week 36. Eligible for the study were women with singleton pregnancy and a fetus in cephalic presentation, admitted for labor, rupture of the membranes or induction after 37 completed gestational weeks. Primigravid women received written information about the study at the maternal health care centers, and eligible women were asked for consent at admission in labor.

Randomization was done at the beginning of the second stage of labor (at full cervical dilatation), in each unit by a telephone call from the delivering midwife to the other department, where randomization lists with numbers for allocation were kept. In women allocated to Ritgen´s maneuver, the protocol stated that the delivery of the fetal head should be managed by this maneuver, i.e. lifting the fetal chin anteriorly, using the fingers of one hand placed between the anus and the coccyx, and thereby extending the fetal neck, whereas the other hand should be placed on the fetal occiput to control the pace of the expulsion of the fetal head. The technique for Ritgen´s maneuver was standardized, and midwives that were unfamiliar with the procedure were instructed by senior colleagues before the trial. In the other study group, the protocol entailed our standard care. The standard practice at delivery was using one hand to apply pressure against the perineum, and the other hand on the fetal occiput to control the expulsion of the fetal head, and only to use Ritgen´s maneuver in case of labor arrest or abnormal fetal heart rate pattern when the fetal head was at the pelvic floor.

ELIGIBILITY:
Inclusion Criteria:

* Women with singleton pregnancy and a fetus in cephalic presentation
* admitted for labor
* rupture of the membranes or induction after 37 completed gestational weeks
* and reaching full cervical dilatation.

Exclusion Criteria:

* Operative delivery

Ages: 16 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1623 (Actual)
Dates: Start 1999-12; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

PRIMARY OUTCOMES:
Perineal rupture grade III-IV (anal sphincter tears) | At delivery - within minutes - hours of randomization

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Herbst, MD, PhD, Principal Investigator — Lund University Hospital
Locations (2):
- Sweden (2):
  - Helsingborgs lasarett, Helsingborg
  - Lund Univeristy Hospital, Lund

REFERENCES:
- [Derived] Jonsson ER, Elfaghi I, Rydhstrom H, Herbst A. Modified Ritgen's maneuver for anal sphincter injury at delivery: a randomized controlled trial. Obstet Gynecol. 2008 Aug;112(2 Pt 1):212-7. doi: 10.1097/AOG.0b013e31817f2867. PMID 18669713